CLINICAL TRIAL: NCT04417959
Title: A Comparison of Visual Functions and Side-effects After DSAEK or DMEK for Fuchs' Endothelial Dystrophy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUH_øjensygdomme_DSAEK_vs_DMEK
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Fuchs' Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Intervention Model Description: Study subjects with the requirement for endothelial keratoplasty and a concomitant need for cataract extraction will be randomized 1:1 to either phaco-DSAEK or phaco-DMEK. Further, a third group consisting of sujects with a solely need for cataract extraction will be included as a control group in our study. The three groups will be prospectively followed.
Who Masked: Participant
Masking Description: Subjects randomized to either phaco-DSAEK or phaco-DMEK will be blinded in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phaco-DSAEK (Other): Subjects randomized to this arm will consist of patients with both Fuchs' endothelial dystrophy and cataract. These will be treated with phacoemulsification and Descemet's stripping automated endothelial keratoplasty.
  Interventions: Procedure: Phaco-DSAEK
- Phaco-DMEK (Other): Subjects randomized to this arm will consist of patients with both Fuchs' endothelial dystrophy and cataract. These will be treated with phacoemulsification and Descemet's membrane endothelial keratoplasty.
  Interventions: Procedure: Phaco-DMEK

INTERVENTIONS:
Procedure: Phaco-DSAEK — The intervention will be performed as a DSAEK triple-procedure with phacoemulsification and intraocular lens implantation prior to DSAEK.
  Arms: Phaco-DSAEK
Procedure: Phaco-DMEK — The intervention will be performed as a DMEK triple-procedure with phacoemulsification and intraocular lens implantation prior to DMEK.
  Arms: Phaco-DMEK

SUMMARY:
Descemet's stripping automated endothelial keratoplasty (DSAEK) and Descemet's membrane endothelial keratoplasty (DMEK) are becoming increasingly popular as treatments for Fuchs' endothelial dystrophy. However, despite several years of use the incidence of cystoid macular edema and damage related to increased intraocular pressure (IOP), and the forward scattering of light through the eye following DSAEK or DMEK have to our knowledge not been prospectively described. Therefore, this project will be a randomized controlled trial investigating these matters.

DETAILED DESCRIPTION:
Purpose:

To investigate 3 different side-effects after DSAEK, DMEK, and cataract extraction (CE) in a randomized controlled trial with 12 months follow-up with CE as an additional control group.

1. To investigate the extend of subclinical cystoid macular edema (CME) and epiretinal membrane (ERM) after DSAEK, DMEK, and CE.
2. To investigate IOP-related changes after DSAEK, DMEK, and CE in means of pupil diameter and cpRNFLT. Further, to describe iris alterations including Urrets-Zavalia Syndrome (UZS).
3. To compare the difference in forward scatter, visual acuity (VA), and low-contrast VA after DSAEK, DMEK, and CE and relate this to the best corrected visual acuity (BCVA). Further, to investigate changes in higher-order aberrations, patient reported outcome measures (PROM), and total corneal refraction after the procedures.

Hypotheses:

1. Subclinical CME and ERM are adverse effects that occur equally often following DSAEK, DMEK, and CE.
2. Following DSAEK, DMEK, and CE, there are no differences in the amount of IOP-related changes in means of pupil diameter,cpRNFLT thinning or iris alterations.
3. Changes in OSI, HOA, PROM, VA, contrast sensitivity, and total corneal refraction occur to the same extend after DSAEK, DMEK, and CE.

Materials and Methods:

Patients referred to the Department of Ophthalmology at Aarhus University Hospital (AUH) for EK or CE will be assessed in order to identify suitable study subjects.

Only patients with primary endothelial failure (Fuchs endothelial dystrophy) and a concomitant need for CE will be considered eligible for randomization to either the DSAEK or the DMEK study groups. Patients included in the study will be randomized 1:1 to the DSAEK or DMEK study groups. Patients referred for CE will be offered to participate in the project and will be included in the CE group. Based on power calculations, it is planned to include 40 patients in each of the 3 groups.

Subject and donor characteristics will be gathered. Subjects with prior uveitis, severe vitreous opacities, diabetes, retinal vein occlusion, glaucoma, age-related macular degeneration, macular atrophy, trauma or corneal grafting will be excluded from the study. Data collection will be conducted at AUH before the interventions and in the follow-up period.

Donor tissue will be prepared in the Danish Cornea Bank, either pre-pealed for DMEK or pre-cut for DSAEK.

Measurements as described below will be conducted both prior to the surgical intervention and 3, 6, and 12 months after this.

Patients lost to follow-up during the project will only be used for analysis at the time-point they have attended. Therefore, for all time-points after the loss to follow-up these subjects will be excluded from our investigation.

In case of capsule rupture where the intraocular lens still is positioned into the lens bag during CE or if rebubbling is needed after DSAEK or DMEK, the subjects will still be eligible for further participation in the project. Adverse events such as primary graft failure or rejection is considered to be rare events for both DSAEK and DMEK and subjects with these will be excluded from our final estimates.

ELIGIBILITY:
Inclusion Criteria:

* Cataract and/or
* Fuch's endothelial dystrophy

Exclusion Criteria:

* Uveitis
* Diabetes mellitus
* Retinal vein occlusion
* Glaucoma
* Exudative age-related macular degeneration
* Advanced macular atrophy
* Ocular trauma
* Prior corneal grafting

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | 12 months
  BCVA will be measured using the early treatment diabetic retinopathy study (ETDRS) chart.

SECONDARY OUTCOMES:
Cystoid macular edema | 3 months
  This will be quantified as central retinal thickness (µm) measured using optical coherence tomography (OCT) scans.
Largest pupil diameter (mm) | 12 months
  The pupil diameter will be measured using the pupillometer DP-2000, Neuroptics.
Iris contraction velocity (mm/s) | 12 months
  The contraction velocity will be measured using the pupillometer DP-2000, Neuroptics.
Circumpapillary Retinal Nerve Fibre Layer Thickness (cpRNFLT) (µm) | 12 months
  The cpRNFLT will be measured using OCT-scans.
Contrast-sensitivity (Weber contrast units) | 12 months
  This will be measured using the Freiburg Visual Acuity and Contrast Test (FrACT)
Forward light scatter | 12 months
  Forward light scatter will be measured using the HD Analyzer, Optical Quality Analysis System (OQAS), Visiometrics. The forward light scatter will be assessed using the objective scattering index (OSI). This system evaluates the intraocular scattering of light.
Higher-order aberrations (HOA) (µm) | 12 months
  Measurements will be performed using Pentacam, Oculus. HOA will be quantified as the root mean square (RMS).

OTHER OUTCOMES:
Epiretinal membrane (ERM) formation | 12 months
  Formation and changes will be assessed using OCT-scans.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Derived] Madsen MBM, Ivarsen A, Hjortdal J. Optical quality after ultrathin Descemet's stripping automated endothelial keratoplasty and Descemet's membrane endothelial keratoplasty: a randomised controlled clinical trial. Br J Ophthalmol. 2025 Dec 11:bjo-2025-328970. doi: 10.1136/bjo-2025-328970. Online ahead of print. PMID 41381122
- [Derived] Madsen MBM, Ivarsen A, Hjortdal J. Visual function after ultrathin Descemet's stripping automated endothelial keratoplasty or Descemet's membrane endothelial keratoplasty combined with cataract surgery: a randomised controlled clinical trial. Br J Ophthalmol. 2024 May 21;108(5):654-661. doi: 10.1136/bjo-2023-323304. PMID 37290822
- [Derived] Molbech Madsen MB, Ivarsen A, Hjortdal J. Macular Thickness After Ultrathin Descemet Stripping Automated Endothelial Keratoplasty and Descemet Membrane Endothelial Keratoplasty Combined With Cataract Surgery: A Randomized Controlled Clinical Trial. Cornea. 2023 Dec 1;42(12):1536-1543. doi: 10.1097/ICO.0000000000003256. Epub 2023 Feb 24. PMID 36853598